CLINICAL TRIAL: NCT03039686
Title: A Randomized, Double Blind, Placebo-Controlled, Study to Assess the Efficacy, Safety, and Tolerability of RO7239361 in Ambulatory Boys With Duchenne Muscular Dystrophy
Brief Title: Clinical Trial to Evaluate the Efficacy, Safety, and Tolerability of RO7239361 in Ambulatory Boys With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN001-016; 2016-001654-18 (EudraCT Number); WN40227 (Other: Hoffman-La Roche)
Record Dates: First submitted 2017-01-27; First posted 2017-02-01 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: muscular dystrophy; Duchenne's Muscular Dystrophy; DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RO7239361 Low Dose (Experimental): Participants received low dose RO7239361 SC on specified days of the 48-week DB period. Following the DB period participants received low dose RO7239361 on specified days for up to 192 weeks during the open-label period followed by 24 weeks of follow-up.
  Interventions: Drug: RO7239361
- RO7239361 High Dose (Experimental): Participants received high dose RO7239361 SC on specified days of the 48-week DB period. Following the DB period participants received high dose RO7239361 on specified days for up to 192 weeks during the open-label period followed by 24 weeks of follow-up.
  Interventions: Drug: RO7239361
- Placebo (Placebo Comparator): Participants received matching placebo solution subcutaneously (SC) on specified days of the 48-week double-blind (DB) period. Following the DB period participants received low dose or high dose RO7239361 on specified days for up to 192 weeks during the open-label period followed by 24 weeks of follow-up.
  Interventions: Drug: Placebo for RO7239361

INTERVENTIONS:
Drug: RO7239361 — Take RO7239361 subcutaneously on specified days over a 48 week blinded period
  Arms: RO7239361 High Dose; RO7239361 Low Dose
Drug: Placebo for RO7239361 — Take placebo subcutaneously on specified days over a 48 week blinded period
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study to assess the efficacy, safety and tolerability of two different weekly doses of RO7239361 in ambulatory boys with Duchenne Muscular Dystrophy (DMD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DMD by confirmed medical history and genetic testing
* Able to walk without assistance
* Minimum North Star Ambulatory Assessment score of 15 at screening
* Able to walk up 4 stairs in 8 seconds or less
* Weigh at least 15 kg (33 lbs)
* Taking corticosteroids for DMD

Exclusion Criteria:

* Any behavior or mental issue that will affect the ability to complete the required study procedures
* Previously or currently taking medications like androgens or human growth hormone
* Use of a ventilator during the day
* Unable to have blood samples collected or receive an injection under the skin
* Concomitant or previous participation at any time in a gene therapy study

Other protocol defined Inclusion/Exclusion Criteria could apply.

Ages: 6 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (44):
- United States (17):
  - Neuromuscular Research Center, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - Yale University School of Medicine ; Pulmonary & Critical Care, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Rush University Medical Center - PPDS, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts Memorial Childrens Medical Center; Department of Neurology, Worcester, Massachusetts
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Las Vegas Clinic, Las Vegas, Nevada
  - Cincinnati Childrens Hospital Medical Center;Investigational Pharmacy, Cincinnati, Ohio
  - Nationwide Childrens Hospital; Research Institute at Nationwide Childrens Hospital, Columbus, Ohio
  - Seattle Children's Hospital, Seattle, Washington
- Instituto centenario, Buenos Aires, Argentina
- Australia (3):
  - Children's Hospital Westmead; Paediatrics & Child Health, Westmead, New South Wales
  - Lady Cilento Children's Hospital; Neurosciences Department, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- UZ Gent, Ghent, Belgium
- Canada (2):
  - London Health Sciences Centre; Children's Hospital; Pediatrics, London, Ontario
  - Children'S Hospital of Eastern Ontario, Ottawa, Ontario
- France (4):
  - Hospices Civils de Lyon, Lyon
  - Hotel Dieu; Service Pharmacie Essais Cliniques, Nantes
  - Hopital Armand Trousseau; centre reference Maladies Neuro-musculaires Est parisien Neuropediatrie, Paris
  - Hopitaux Universitaires de Strasbourg, Strasbourg
- Universitatsklinikum Essen; Innere Klinik, Essen, Germany
- Italy (3):
  - Fondazione Serena Onlus - CENTRO CLINICO NEMO, Milano, Emilia-Romagna
  - Fondazione Policlinico Universitario A Gemelli; Servizio di Farmacia, Rome, Lazio
  - Az. Osp. Universitaria Pol. G. Martino; Dip. Neuroscienze, Scienze Psichiatriche e Anest., Messina, Sicily
- Japan (5):
  - Hyogo College of Medicine Hospital, Hyōgo
  - Miyagi Children's Hospital, Miyagi
  - Shinshu University Hospital, Nagano
  - National Hospital Organization Osaka Toneyama Medical Center, Osaka
  - National Center of Neurology and Psychiatry, Tokyo
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud University Nijmegen Medical Centre; Ophthalmology, Nijmegen
- Spain (2):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital Universitari i Politecnic La Fe de Valencia; Servicio de Farmacia, Valencia
- Drottning Silvias Barn- och ungdomssjukhus; Kliniken for barnmedicin, Gothenburg, Sweden
- United Kingdom (2):
  - Alder Hey Children s Hospital; Department of Pediatrics, Liverpool
  - UCL Institute of Child Health & Great Ormond Street Hospital for Children, London

REFERENCES:
- [Derived] Muntoni F, Byrne BJ, McMillan HJ, Ryan MM, Wong BL, Dukart J, Bansal A, Cosson V, Dreghici R, Guridi M, Rabbia M, Staunton H, Tirucherai GS, Yen K, Yuan X, Wagner KR; Taldefgrobep Alfa Study Group. The Clinical Development of Taldefgrobep Alfa: An Anti-Myostatin Adnectin for the Treatment of Duchenne Muscular Dystrophy. Neurol Ther. 2024 Feb;13(1):183-219. doi: 10.1007/s40120-023-00570-w. Epub 2024 Jan 8. PMID 38190001
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Provides information about the Roche clinical trial NCT03039686 and molecule being investigated in Duchenne — http://roche-duchenne-clinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Double-blind Period
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Started | 56 | 55 | 55
Completed | 29 | 26 | 32
Not Completed | 27 | 29 | 23
Not completed — Administrative Reason by Sponsor | 24 | 25 | 21
Not completed — Subject Request to Discontinue Study Treatment | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Death | 0 | 0 | 1
Period: Open Label Period
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Started | 0 (Double-blind (DB) placebo participants switched to RO7239361 (RO) for the open label phase.) | 38 (14 DB placebo participants switched to the RO Low Dose for the open-label phase.) | 42 (13 DB placebo participants switched to the RO High Dose for the open-label phase.)
Completed DB, Did Not Start OL | 2 | 2 | 3
Completed | 0 | 0 | 0
Not Completed | 0 | 38 | 42
Not completed — Administrative Reason by Sponsor | 0 | 34 | 41
Not completed — Subject Request to Discontinue Study Treatment | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose | Total
Number analyzed (Participants) | 56 | 55 | 55 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (1.7) | 8.5 (1.8) | 8.4 (1.5) | 8.5 (1.7)
Age, Customized [Number; unit: participants]
  Children (6-11 years) | 56 | 55 | 55 | 166
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 56 | 55 | 55 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 6 | 18
  Not Hispanic or Latino | 43 | 41 | 43 | 127
  Unknown or Not Reported | 6 | 9 | 6 | 21
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 9 | 7 | 7 | 23
  Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 1
  White | 42 | 45 | 45 | 132
  Other | 5 | 3 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Baseline for the North Star Ambulatory Assessment (NSAA) Total Score
Description: The NSAA is a functional scale specifically designed for ambulant boys with Duchenne muscular dystrophy (DMD) that can provide information about motor function. The NSAA is a 17-item test of standing, ability to transition from lying to sitting, sitting to standing, and other mobility assessments. Each of the 17 items is evaluated on an ordinal scale of 0-2: 0 = unable to achieve independently, 1 = modified method but achieves goal independent of physical assistance from another, or 2 = normal with no obvious modification of activity. Total score range is 0 to 34. Higher scores reflect better performance.
Time Frame: Baseline
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
score on a scale | 23.1 (6.4) | 24.5 (5.5) | 22.7 (6.7)

2. Primary Outcome: Change From Baseline in the North Star Ambulatory Assessment (NSAA) Total Score at Week 48
Description: The NSAA is a functional scale specifically designed for ambulant boys with Duchenne muscular dystrophy (DMD) that can provide information about motor function. The NSAA is a 17-item test of standing, ability to transition from lying to sitting, sitting to standing, and other mobility assessments. Each of the 17 items is evaluated on an ordinal scale of 0-2: 0 = unable to achieve independently, 1 = modified method but achieves goal independent of physical assistance from another, or 2 = normal with no obvious modification of activity. Total score range is 0 to 34. Higher scores reflect better performance. A positive change from baseline indicates an improvement. Based on the mixed-effect model of repeated measures (MMRM).
Time Frame: Baseline, Week 48
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment. MMRM analysis included all participants at baseline and the following number of participants by Week 48: Placebo n=30, Low Dose n=29, High Dose n=33.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
score on a scale | -2.99 (0.65) | -3.44 (0.67) | -2.41 (0.64)
Statistical Analysis 1: Comparison: Placebo vs RO7239361 Low Dose; Test type: Superiority; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-2.17 to 1.27], Standard Error of Mean 0.87 — Based on the MMRM using an unstructured covariance matrix -change = Baseline + Age Interactive response system (IXRS) Stratum + Corticosteroid Regimen IXRS Stratum + Analysis Visit*Treatment
Statistical Analysis 2: Comparison: Placebo vs RO7239361 High Dose; Test type: Superiority; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-1.10 to 2.26], Standard Error of Mean 0.85 — Based on the MMRM using an unstructured covariance matrix -change = Baseline + Age IXRS Stratum + Corticosteroid Regimen IXRS Stratum + Analysis Visit*Treatment

3. Secondary Outcome: Baseline Time for 4 Stair Climb
Description: The time to complete the 4 stair climb was measured at baseline.
Time Frame: Baseline
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment.
Measure: Mean (Standard Deviation); unit: seconds (secs)
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
seconds (secs) | 3.81 (1.55) | 3.85 (1.61) | 3.92 (1.91)

4. Secondary Outcome: Change From Baseline at Week 48 in 4 Stair Climb Velocity (4SCV)
Description: 4SCV was calculated as the ratio of the number of stairs climbed (4) divided by the number of seconds taken to complete the 4-stair climb. The results were converted into velocity (distance/time). A positive change from baseline indicates an improvement. Based on the mixed-effect model of repeated measures (MMRM).
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: stairs/sec
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
stairs/sec | -0.15 (0.07) | -0.15 (0.07) | -0.07 (0.07)
Statistical Analysis 1: Comparison: Placebo vs RO7239361 Low Dose; Test type: Superiority; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.21 to 0.20], Standard Error of Mean 0.10 — Based on the MMRM using an unstructured covariance matrix - change = Baseline + Age IXRS Stratum + Corticosteroid Regimen IXRS Stratum + Analysis Visit*Treatment
Statistical Analysis 2: Comparison: Placebo vs RO7239361 High Dose; Test type: Superiority; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.12 to 0.27], Standard Error of Mean 0.10 — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Baseline for the Time to Stand From Supine
Description: The time required for a participant to stand from supine position. A longer time reflects a worse outcome.
Time Frame: Baseline
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment.
Measure: Mean (Standard Deviation); unit: secs
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
secs | 6.28 (4.75) | 6.15 (4.07) | 7.24 (9.22)

6. Secondary Outcome: Change From Baseline at Week 48 in Stand From Supine Velocity
Description: The time required for a participant to stand from supine position. A longer time reflects a worse outcome. A negative change from baseline indicates an improvement. Based on the mixed-effect model of repeated measures (MMRM).
Time Frame: Baseline, Week 48
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment. MMRM analysis included all participants at baseline and the following number of participants by Week 48: Placebo n=28, Low Dose n=28, High Dose n=32.
Measure: Least Squares Mean (Standard Error); unit: 1/sec
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
1/sec | -0.05 (0.01) | -0.02 (0.01) | -0.02 (0.01)
Statistical Analysis 1: Comparison: Placebo vs RO7239361 Low Dose; Test type: Superiority; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.00 to 0.06], Standard Error of Mean 0.02 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RO7239361 High Dose; Test type: Superiority; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.00 to 0.06], Standard Error of Mean 0.02 — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Baseline Time for 10 Meter Walk/Run
Description: The time required for a participant to run or walk a distance of 10 meters as quickly as possible. A longer time reflects a worse outcome.
Time Frame: Baseline
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment.
Measure: Mean (Standard Deviation); unit: secs
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
secs | 5.38 (1.48) | 5.51 (1.68) | 5.68 (2.30)

8. Secondary Outcome: Change From Baseline at Week 48 in 10 M Walk/Run Velocity
Description: The time required for a participant to run or walk a distance of 10 meters as quickly as possible calculated as velocity (distance/time). A positive change from baseline indicates an improvement. Based on the mixed-effect model of repeated measures (MMRM).
Time Frame: Baseline, Week 48
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment. MMRM analysis included all participants at baseline and the following number of participants by Week 48: Placebo n=30, Low Dose n=29, High Dose n=31.
Measure: Least Squares Mean (Standard Error); unit: m/sec
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
m/sec | -0.23 (0.06) | -0.14 (0.07) | -0.23 (0.06)
Statistical Analysis 1: Comparison: Placebo vs RO7239361 Low Dose; Test type: Superiority; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.08 to 0.27], Standard Error of Mean 0.09 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RO7239361 High Dose; Test type: Superiority; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.17 to 0.18], Standard Error of Mean 0.09 — [estimate comment as in outcome 4, analysis 1]

9. Secondary Outcome: Baseline for the Pediatric Outcome Data Collection Instrument (PODCI) Transfer and Basic Mobility Subscale
Description: The PODCI is designed to be completed by the parent/guardian of a child who has knowledge of the child's conditions. The Transfer and Basic Mobility scale is one of the subscales of the PODCI. The results are standardized into a scale of 0-100 with a higher score reflecting better performance.
Time Frame: Baseline
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
score on a scale | 85.59 (10.21) | 86.54 (9.52) | 84.47 (14.76)

10. Secondary Outcome: Change From Baseline at Week 48 in Pediatric Outcome Data Collection Instrument (PODCI) Transfer and Basic Mobility Subscale
Description: The PODCI is designed to be completed by the parent/guardian of a child who has knowledge of the child's conditions. The Transfer and Basic Mobility scale is one of the subscales of the PODCI. The results are standardized into a scale of 0-100 with a higher score reflecting better performance. A positive change from baseline indicates an improvement. Based on the mixed-effect model of repeated measures (MMRM).
Time Frame: Baseline, Week 48
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment. MMRM analysis included all participants at baseline and the following number of participants by Week 48: Placebo n=31, Low Dose n=29, High Dose n=34.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
score on a scale | -5.47 (1.79) | -7.47 (1.83) | -4.51 (1.77)
Statistical Analysis 1: Comparison: Placebo vs RO7239361 Low Dose; Test type: Superiority; Mean Difference (Final Values) = -2.00, 95% CI 2-sided [-6.76 to 2.77], Standard Error of Mean 2.41 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RO7239361 High Dose; Test type: Superiority; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-3.71 to 5.63], Standard Error of Mean 2.36 — [estimate comment as in outcome 4, analysis 1]

11. Secondary Outcome: Change From Baseline at Week 48 in Proximal Lower Extremity Flexor Strength
Description: Proximal lower extremity flexor (knee extension and knee flexion) strength was measured using manual myometry. A higher score reflects a better outcome. A positive change from baseline indicates an improvement.
Time Frame: Baseline, Week 48
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
kilogram (kg)
  Baseline: Knee Extenders: number analyzed (Participants) | 56 | 55 | 54
  Baseline: Knee Extenders | 5.58 (2.87) | 6.25 (3.63) | 5.76 (3.53)
  Change from Baseline at Week 48: Knee Extenders: number analyzed (Participants) | 30 | 28 | 33
  Change from Baseline at Week 48: Knee Extenders | -1.19 (2.13) | -0.47 (2.43) | -0.88 (2.97)
  Baseline: Knee Flexors: number analyzed (Participants) | 56 | 55 | 54
  Baseline: Knee Flexors | 5.04 (2.58) | 5.70 (3.08) | 5.04 (2.72)
  Change from Baseline at Week 48: Knee Flexors: number analyzed (Participants) | 30 | 28 | 33
  Change from Baseline at Week 48: Knee Flexors | 0.15 (2.24) | 0.08 (2.53) | -0.13 (2.29)

12. Secondary Outcome: Baseline for the 6 Minute Walk Distance (6MWD)
Description: The 6MWD measured the distance a participant was able to traverse while walking for 6 minutes. A longer distance reflects a better outcome.
Time Frame: Baseline
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment.
Measure: Mean (Standard Deviation); unit: meters (m)
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
meters (m) | 388.33 (69.59) | 399.73 (68.35) | 370.73 (93.35)

13. Secondary Outcome: Change From Baseline at Week 48 in 6 Minute Walk Distance (6MWD)
Description: The 6MWD measured the distance a participant was able to traverse while walking for 6 minutes. A longer distance reflects a better outcome. A positive change from baseline indicates an improvement. Based on the mixed-effect model of repeated measures (MMRM).
Time Frame: Baseline, Week 48
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment. MMRM analysis included all participants at baseline and the following number of participants by Week 48: Placebo n=29, Low Dose n=25, High Dose n=31.
Measure: Least Squares Mean (Standard Error); unit: meters (m)
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55
meters (m) | -41.3 (8.7) | -39.6 (9.0) | -30.0 (8.7)
Statistical Analysis 1: Comparison: Placebo vs RO7239361 Low Dose; Test type: Superiority; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-21.1 to 24.6], Standard Error of Mean 11.5 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RO7239361 High Dose; Test type: Superiority; Mean Difference (Final Values) = 11.3, 95% CI 2-sided [-11.0 to 33.6], Standard Error of Mean 11.3 — [estimate comment as in outcome 4, analysis 1]

14. Secondary Outcome: Percentage of Participants for Each Clinical Global Impression of Change (CGI-C) Assessment Status at Week 48
Description: The CGI-C was used to assess the participant's overall condition on a 7-point scale, using the status markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse or very much worse" at Week 48 as compared to baseline.
Time Frame: Baseline, Week 48
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment. Included in the analysis are only those subjects for whom an efficacy assessment was completed at Week 48.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 36 | 37 | 31
percentage of participants
  Very much improved | 0 | 0 | 0
  Much improved | 5.6 | 2.7 | 3.2
  Minimally improved | 13.9 | 13.5 | 19.4
  No change | 58.3 | 54.1 | 51.6
  Minimally worse | 16.7 | 18.9 | 22.6
  Much worse | 5.6 | 10.8 | 3.2
  Very much worse | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline at Week 48 in 95th Percentile Stride Velocity
Description: Stride velocity was recorded with the ActiMyo device in a subset of the overall study population. The ActiMyo device measures the daily movement and activity levels of the participant. The device consists of two sensors worn on each ankle. A higher velocity reflects a better outcome. A positive change from baseline indicates an improvement.
Time Frame: Baseline, Week 48
Population: Intent-to-Treat (ITT) population included all enrolled participants who received a randomization treatment assignment.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Placebo | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 17 | 19 | 15
m/sec
  Baseline | 1.69 (0.33) | 1.54 (0.35) | 1.57 (0.46)
  Change from Baseline at Week 48: number analyzed (Participants) | 5 | 7 | 4
  Change from Baseline at Week 48 | -0.25 (0.39) | -0.22 (0.22) | -0.28 (0.29)

16. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: During DB period (48 weeks) and Whole study (up to approximately 34 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study therapy. Data are presented for the arms in the DB period as well as for all RO7239361-treated participants in the whole study.
Measure: Number; unit: participants
Groups:
- Placebo DB: Participants received matching placebo solution subcutaneously (SC) on specified days of the 48-week double-blind (DB) period.
- RO7239361 Low Dose DB: Participants received low dose RO7239361 SC on specified days of the 48-week DB period.
- RO7239361 High Dose DB: Participants received high dose RO7239361 SC on specified days of the 48-week DB period.
- RO7239361 High Dose Whole Study: Participants received high dose SC on specified days of the 48-week DB period. Following the DB period participants received high dose RO7239361 on specified days for up to 192 weeks during the open-label period followed by 24 weeks of follow-up.
Arm/Group | Placebo DB | RO7239361 Low Dose DB | RO7239361 High Dose DB | RO7239361 Low Dose | RO7239361 High Dose Whole Study
Number analyzed (Participants) | 56 | 55 | 55 | 69 | 68
participants
  Double-Blind Period: number analyzed (Participants) | 56 | 55 | 55 | 0 | 0
  Double-Blind Period | 46 | 48 | 49 |  |
  Whole Study: number analyzed (Participants) | 0 | 0 | 0 | 69 | 68
  Whole Study |  |  |  | 57 | 56

17. Secondary Outcome: Number of Participants With AEs Leading to Discontinuation
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. Reported here is the number of participants with AEs that led to study discontinuation.
Time Frame: During DB period (48 weeks) and Whole study (up to approximately 34 months)
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Placebo DB | RO7239361 Low Dose DB | RO7239361 High Dose DB | RO7239361 Low Dose | RO7239361 High Dose
Number analyzed (Participants) | 56 | 55 | 55 | 69 | 68
participants
  Double-Blind Period: number analyzed (Participants) | 56 | 55 | 55 | 0 | 0
  Double-Blind Period | 0 | 0 | 0 |  |
  Whole Study: number analyzed (Participants) | 0 | 0 | 0 | 69 | 68
  Whole Study |  |  |  | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 34 months
Description: Safety population included all enrolled participants who received at least 1 dose of study therapy.
Groups:
- Placebo, Then RO7239361 Low Dose OL: Participants received matching placebo solution SC on specified days of the 48-week DB period. Following the DB period participants received low dose RO7239361 on specified days for up to 192 weeks during the open-label (OL) period followed by 24 weeks of follow-up.
- Placebo, Then RO7239361 High Dose OL: Participants received matching placebo solution SC on specified days of the 48-week DB period. Following the DB period participants received high dose RO7239361 on specified days for up to 192 weeks during the open-label period followed by 24 weeks of follow-up.
- RO7239361 Low Dose, Then RO7239361 Low Dose OL: Participants received low dose RO7239361 SC on specified days of the 48-week DB period. Following the DB period participants received low dose RO7239361 on specified days for up to 192 weeks during the open-label period followed by 24 weeks of follow-up.
- RO7239361 High Dose, Then RO7239361 High Dose OL: Participants received high dose RO7239361 SC on specified days of the 48-week DB period. Following the DB period participants received high dose RO7239361 on specified days for up to 192 weeks during the open-label period followed by 24 weeks of follow-up
Arm/Group | Placebo DB | RO7239361 Low Dose DB | RO7239361 High Dose DB | Placebo, Then RO7239361 Low Dose OL | Placebo, Then RO7239361 High Dose OL | RO7239361 Low Dose, Then RO7239361 Low Dose OL | RO7239361 High Dose, Then RO7239361 High Dose OL
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/55 | 1/55 | 0/14 | 0/13 | 0/24 | 0/29
Serious Adverse Events (participants affected / at risk) | 3/56 | 2/55 | 4/55 | 0/14 | 0/13 | 0/24 | 0/29
Other Adverse Events (participants affected / at risk) | 43/56 | 43/55 | 47/55 | 8/14 | 7/13 | 13/24 | 12/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo DB (N=56) | RO7239361 Low Dose DB (N=55) | RO7239361 High Dose DB (N=55) | Placebo, Then RO7239361 Low Dose OL (N=14) | Placebo, Then RO7239361 High Dose OL (N=13) | RO7239361 Low Dose, Then RO7239361 Low Dose OL (N=24) | RO7239361 High Dose, Then RO7239361 High Dose OL (N=29)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo DB (N=56) | RO7239361 Low Dose DB (N=55) | RO7239361 High Dose DB (N=55) | Placebo, Then RO7239361 Low Dose OL (N=14) | Placebo, Then RO7239361 High Dose OL (N=13) | RO7239361 Low Dose, Then RO7239361 Low Dose OL (N=24) | RO7239361 High Dose, Then RO7239361 High Dose OL (N=29)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 4 (5) | 7 (12) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Constipation (Gastrointestinal disorders) | 4 (5) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 10 (13) | 4 (8) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (9) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 6 (6) | 8 (14) | 6 (11) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Fatigue (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gait inability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 2 (3) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 8 (25) | 11 (43) | 12 (38) | 0 (0) | 3 (17) | 2 (6) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 3 (7) | 2 (9) | 1 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 2 (2) | 2 (6) | 0 (0) | 1 (12) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (3) | 4 (29) | 2 (33) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 4 (31) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (8) | 9 (13) | 8 (9) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 13 (17) | 13 (17) | 13 (16) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 3 (5) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (8) | 4 (5) | 7 (16) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 5 (7) | 4 (5) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 5 (11) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gadolinium deposition disease (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 4 (4) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (3) | 3 (12) | 0 (0) | 1 (3) | 0 (0) | 1 (4) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glutamate dehydrogenase increased (Investigations) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (8) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (7) | 2 (6) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (6) | 8 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 9 (28) | 14 (60) | 10 (42) | 1 (3) | 0 (0) | 2 (9) | 2 (4)
Migraine (Nervous system disorders) | 0 (0) | 1 (10) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (11) | 7 (13) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (9) | 3 (15) | 6 (17) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (9) | 4 (5) | 7 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT03039686/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT03039686/SAP_001.pdf